CLINICAL TRIAL: NCT06559735
Title: A Prospective, Observational Study Examining Local Cerebral Oxygenation in Chronic Pain Patients Utilizing Spinal Cord Stimulation
Brief Title: Local Cerebral Oxygenation in Chronic Pain Patients Utilizing Spinal Cord Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CereVu Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CIP-5005
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SCS Study Arm (Experimental): Within subject observational arm measuring non-invasive cerebral oxygenation/flow before, during and after SCS.
  Interventions: Device: CereVu Device

INTERVENTIONS:
Device: CereVu Device — Observational, non-invasive measurements

SUMMARY:
The primary objective of the study is to determine changes in cerebral nociceptive hemodynamic response (blood oxygenation/flow) before, during and following spinal cord stimulation (SCS). Objective measurements of cerebral nociceptive hemodynamic responses will be obtained with the CereVu sensor and ROPA system and will be analyzed offline and compared against subjective measures of pain. Proprietary analysis algorithms will be incorporated and developed to understand how the objective measurements correlate with subject reported pain levels

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older at the time of enrolment
2. Diagnosed with chronic, intractable pain of the trunk and/or limbs, which has been refractory to conservative therapy for a minimum of 6 months
3. Subject has a minimum Visual Analog Scale (VAS) score of 50 mm or higher (where 100 mm indicates the worst imaginable pain) at baseline or a 5 on a Numerical Rating Scale (NRS)
4. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician
5. Be willing and capable of giving informed consent
6. Be willing and able to comply with study-related requirements, procedures, and visits

Exclusion Criteria:

1. Subject is pregnant or nursing
2. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, as determined by the Investigator
3. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention, and/or ability to evaluate treatment outcomes
4. Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker, deep brain stimulator (DBS), or sacral nerve stimulator (SNS)
5. Have prior experience with SCS
6. Be concomitantly participating in another clinical study
7. Subject has secondary gain issues that could interfere with the study measures or outcomes
8. Subject is contraindicated for use of non-invasive cerebral oxygenation measurements (e.g., at risk for sensor displacement such as facial cosmetic. Non-intact skin on the forehead, or ENT surgery)
9. Subject is allergic to any adhesives, materials or fluids in or used in conjunction with the CereVu sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Regional Cerebral Oxygenation/Blood Flow | 1 week
  Opital Spectophotometry measurement from the forehead
Numerical Pain Rating Scale (NRS) | 1 week
  Subjective pain 11-point pain scale

SECONDARY OUTCOMES:
Stress/Anxiety | 1 week
  Hamilton Anxiety Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jon Gasson, Study Director — CereVu
Locations (1):
- Boomerang Healthcare, Walnut Creek, California, United States

IPD SHARING:
Plan to Share IPD: No